CLINICAL TRIAL: NCT04222673
Title: Evaluating the Use of Peer Specialists to Support Suicide Prevention
Brief Title: Peer Based Suicide Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: D3291-P; RX003291-01A1 (Other Grant/Funding Number: Office of Research & Development)
Record Dates: First submitted 2020-01-03; First posted 2020-01-10 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Suicide
Keywords: Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: The intervention will last 3-months, a time frame that overlaps with the typical duration of a VA suicide high risk flag. Meetings will be 30-45 minutes and occur primarily in the community, home, or by telephone. Session content will be rooted in Peer Specialists (PSs) offering nonjudgmental empathic support, active listening, and constructive disclosure and role modeling. A primary focus will be helping patients with flags to identify and strengthen connections with informal supports and participation in activities in their community that will enable them to feel more worthwhile as individuals and hopeful about their future.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peer Specialist (Experimental): The intervention will last 3-months, a time frame that overlaps with the typical duration of a VA suicide high risk flag. Meetings will be 30-45 minutes and occur primarily in the community, home, or by telephone. Session content will be rooted in Peer Specialists (PSs) offering nonjudgmental empathic support, active listening, and constructive disclosure and role modeling. A primary focus will be helping patients with flags to identify and strengthen connections with informal supports and participation in activities in their community that will enable them to feel more worthwhile as individuals and hopeful about their future.
  Interventions: Behavioral: Peer Specialist Suicide Prevention

INTERVENTIONS:
Behavioral: Peer Specialist Suicide Prevention — The intervention will last 3-months, a time frame that overlaps with the typical duration of a VA suicide high risk flag. Meetings will be 30-45 minutes and occur primarily in the community, home, or by telephone. Session content will be rooted in Peer Specialists (PSs) offering nonjudgmental empathic support, active listening, and constructive disclosure and role modeling. A primary focus will be helping patients with flags to identify and strengthen connections with informal supports and participation in activities in their community that will enable them to feel more worthwhile as individuals and hopeful about their future.

SUMMARY:
Veterans Health Administration (VHA) suicide rates remain high, requiring new approaches. VHA patients tend to have high medical and behavioral health care needs that cause disruption in their lives and heighten their risk of suicide. This study will adapt and pilot test an intervention that expands the focus of care for VHA patients with high risk for suicide to building a life of self-respect, meaning, and connectedness in one's local community. The pilot intervention will involve receiving support and mentorship from a fellow Veteran living with the same challenges who has been trained in helping others manage their disabilities while achieving specific life goals (i.e., a 'Peer Specialist'). Results from this study will demonstrate the preliminary effectiveness of supplementing the VHA's current clinical approaches to suicide prevention with support provided by a trained Peer Specialist that offers empathy, hope, and practical advice that stemming from 'lived experience' of disability and recovery.

DETAILED DESCRIPTION:
The investigators have assembled a team of clinical psychologists and researchers to use Intervention Mapping (IM) to adapt and test PREVAIL (a non VA, peer specialist based suicide prevention program) as a Peer Specialist (PS)-delivered intervention to reduce suicide ideation in VA patients who are at high risk of suicide. Building on the investigators' work with PSs, suicide research, and participatory methods, the investigators will begin the IM process with a needs assessment that includes interviews with PSs, VHA patients, providers, and directors (n=12) to assess attitudes and perceptions of current clinical practices for high risk Veterans, PSs, and areas of possible improvement in suicide prevention. This information will be shared with a steering committee to begin adapting PREVAIL to patients with high suicide risk in VHA. Following best practices for pilot investigations and intervention adaptation, the investigators will recruit 12 VHA patients with unipolar or bipolar depression flagged for high suicide risk to participate in a "pre-pilot" and provide feedback on how the adapted intervention may be revised. After making any necessary modifications to the intervention, the investigators will recruit a second group of 12 high risk Veterans for a "formal pilot" to further evaluate the feasibility and acceptability of recruitment, retention, and assessment procedures for a large randomized trial. Outcome variables will include health care visits for suicide-related reasons and self-reported suicidal ideation/acts as well as several outcomes that are rehabilitative in nature, such as self-rated community integration; sense of hope, meaning, and purpose; and self-esteem and social support. The investigators aim to: Aim 1: Use Intervention Mapping to identify which components of PREVAIL require adaptation to reduce suicidal ideation in high risk VHA patients and to identify implementation strategies in the VHA system; Aim 2: Pilot test the feasibility and acceptability of the adapted PREVAIL, rehabilitative measures, and suicide-related outcomes for use in a rigorous prospective study.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will target Veterans with suicide flags because they are at greatest risk for suicide and therefore most in need of intervention
* Eligibility will be limited to Veterans diagnosed with unipolar or bipolar depression as this diagnostic group is the most prevalent in suicidal samples and is supported by prior meta-analyses on peer-provided interventions
* The investigators will ensure decision-making capacity using the Blessed Orientation, Memory, Concentration Test and a brief quiz about the study
* This quiz will involve an iterative process of querying the participants' understanding of consent information with a 10-item true/false test and providing feedback until an acceptable level of understanding is achieved (must get 100% correct after 3 tries to enroll)

Exclusion Criteria:

* cognitive impairment as indicated by a Blessed score of >10
* unable to provide voluntary, written informed consent for any reason

  * e.g., incompetency
* determination by the patient's psychiatrist not to be appropriate for participation due to unstable psychosis, cognitive disorder, or severe personality disorder
* residing more than 50 miles away

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Chinman, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (3):
- United States (3):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schmutte T, Krishnamurti LS, Davidson L, Klee A, Bullock J, Panas RM, Pfeiffer PN, Chinman M. Implementing Peer Specialists in Suicide Prevention Efforts in the Veterans Health Administration. Psychiatr Q. 2023 Jun;94(2):311-319. doi: 10.1007/s11126-023-10034-x. Epub 2023 Jun 6. PMID 37278930

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Given the nature of the subject matter (suicide), recruitment for the study was extremely challenging. Therefore, instead of having a pre-pilot and then a formal pilot, we collected data all at once in one pilot. That is why we are reporting the data all together in one group.
  Also, the 'needs assessment' process was simply informal qualitative discussions with various stakeholders that helped us adapt the programs to the VA. That is why the information is not reported here.
Period: Overall Study
Arm/Group | Peer Specialist
Started | 17
Completed | 12
Not Completed | 5
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Population: Only baseline data for 12 individuals was reported because the 5 who dropped out left very quickly, so quickly that they did not feel like they were even part of the study.
Arm/Group | Peer Specialist
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Questionnaire About the Process of Recovery (QPR) Change
Description: The Questionnaire about the Process of Recovery (QPR), contains 15 items that measure connectedness, hope, identity, meaning, and empowerment. The QPR has demonstrated high internal and convergent validity as well as sensitivity to change. Range=0-60. High scores reflect greater connectedness, hope, positive identify, meaning, and empowerment.
Time Frame: Baseline, post intervention (12 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Peer Specialist: 3 month PREVAIL intervention
Arm/Group | Peer Specialist
Number analyzed (Participants) | 12
score on a scale
  Baseline | 48.3 (10.9)
  Post | 50.1 (11.9)
Statistical Analysis 1: Comparison: Peer Specialist; Test type: Superiority — Given the small sample size and recommendations for pilot studies, quantitative analyses were descriptive (frequencies, means) and based on the Reliable Change Index (RCI) for each participant for each outcome measure. The RCI is used to determine whether pre- to post- score differences are statistically reliable and to categorize changes as either improved, deteriorated, or indeterminate. A statistical threshold of RCI score z = + 1.96 and p < .05 was used to establish clinical significance; p = .05, the Reliable Change Index

2. Primary Outcome: Hearth Hope Index
Description: a 12-item index shown to be reliable (a=.97) and valid, correlating with the Existential Well-Being Scale (r=.84) and the Hopelessness Scale (r=-.73). Scoring consists of summing the points for each item (ranges from 1 - least amount of hope to 4, indicating the most amount of hope) to make a total scale. Total possible points on the total scale is 48 points; the lowest is 12. The higher the score the higher the level of hope.
Time Frame: Baseline, post intervention (12 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer Specialist
Number analyzed (Participants) | 12
score on a scale
  Baseline | 27.5 (6.84)
  Post | 29.2 (7.93)
Statistical Analysis 1: Comparison: Peer Specialist; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .05, the Reliable Change Index

3. Primary Outcome: Suicide Cognitions Scale (SCS) Change
Description: The Suicide Cognitions Scale (SCS), contains18 items that assess thoughts of unlovability, unsolvability, and unbearability. The SCS has strong psychometric qualities in diverse samples (including Veterans) with incremental validity to predicting suicidal behavior beyond depression, INQ scores, prior attempts, and suicidal ideation. Range 18-90. Higher scores reflected greater sense of unlovability and inability to cope
Time Frame: Baseline, post intervention (12 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer Specialist
Number analyzed (Participants) | 12
score on a scale
  Baseline | 38.8 (7.78)
  Post | 36.3 (11.2)
Statistical Analysis 1: Comparison: Peer Specialist; Given the small sample size and recommendations for pilot studies, quantitative analyses were descriptive (frequencies, means) and based on the Reliable Change Index (RCI) for each participant for each outcome measure. The RCI is used to determine whether pre- to post- score differences are statistically reliable and to categorize changes as either improved, deteriorated, or indeterminate. A statistical threshold of RCI score z = + 1.96 and p < .05 was used to establish clinical significance; Test type: Other; p = .05, the Reliable Change Index

4. Primary Outcome: Interpersonal Needs Questionnaire (INQ) Change - Perceived Burden
Description: The Interpersonal Needs Questionnaire (INQ) uses 15 items to measure two underlying motives for suicidal desire (i.e., perceived burden and thwarted belonging). The INQ has established validity and reliability, including with on Veterans. Range 15-105. Higher scores associated with greater sense of perceived burden and thwarted belongingness.
Time Frame: Baseline, post intervention (12 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer Specialist
Number analyzed (Participants) | 12
score on a scale
  Baseline | 20.7 (9.56)
  Post | 20.3 (11.7)
Statistical Analysis 1: Comparison: Peer Specialist; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = .05, the Reliable Change Index

5. Primary Outcome: Interpersonal Needs Questionnaire (INQ) Change - Thwarted Belonging
Description: as for outcome 4
Time Frame: Baseline, post intervention (12 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer Specialist
Number analyzed (Participants) | 12
score on a scale
  Baseline | 37.3 (7.02)
  Post | 41.1 (8.86)
Statistical Analysis 1: Comparison: Peer Specialist; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = .05, the Reliable Change Index

6. Primary Outcome: Quick Inventory of Depressive Symptoms (QIDS) Change
Description: To assess depression symptoms, the investigators will use the Quick Inventory of Depressive Symptoms (QIDS) which consists of 16 questions to assess depression severity. The QIDS has demonstrated high reliability, validity, and sensitivity to treatment change, including among Veterans. Range=0-27. Higher scores represent increasing severity of depression.
Time Frame: Baseline, post intervention (12 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer Specialist
Number analyzed (Participants) | 12
score on a scale
  Baseline | 19.4 (8.51)
  Post | 17.3 (8.34)
Statistical Analysis 1: Comparison: Peer Specialist; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .05, the Reliable Change Index

7. Primary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS) - Suicidal Ideation
Description: Suicide measures will include the Columbia-Suicide Severity Rating Scale (C-SSRS) to assess suicidal ideation (past 30 days) and behaviors (past 3 months). Suicide ideation items include: (1) wish to be dead, (2) nonspecific active suicidal thoughts, (3) suicidal thoughts with methods, (4) suicidal intent, and (5) suicidal intent with plan. The suicidal behavior subscales include: (1) attempts (actual, aborted interrupted), (2) preparatory behavior, and (3) non-suicidal self-injurious behavior. Range= 0-10. Higher scores represent increasing presence of suicide-related behaviors and thoughts.
Time Frame: Baseline, post intervention (12 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer Specialist
Number analyzed (Participants) | 12
score on a scale
  Baseline | 2.67 (1.78)
  Post | 1.08 (.99)
Statistical Analysis 1: Comparison: Peer Specialist; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = .05, the Reliable Change Index

8. Primary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS) - Suicidal Ideation Intensity
Description: Suicide measures will include the Columbia-Suicide Severity Rating Scale (C-SSRS) to assess suicidal ideation (past 30 days) and behaviors (past 3 months). Suicide ideation items include: (1) wish to be dead, (2) nonspecific active suicidal thoughts, (3) suicidal thoughts with methods, (4) suicidal intent, and (5) suicidal intent with plan. The suicidal behavior subscales include: (1) attempts (actual, aborted interrupted), (2) preparatory behavior, and (3) non-suicidal self-injurious behavior. Range= 0-25. Higher scores represent increasing presence of suicide-related behaviors and thoughts.
Time Frame: Baseline, post intervention (12 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer Specialist
Number analyzed (Participants) | 12
score on a scale
  Baseline | 11.8 (4.99)
  Post | 9.42 (7.69)
Statistical Analysis 1: Comparison: Peer Specialist; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = .05, the Reliable Change Index

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Peer Specialist
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT04222673/Prot_001.pdf
  • Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT04222673/SAP_002.pdf
  • Informed Consent Form (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT04222673/ICF_000.pdf